CLINICAL TRIAL: NCT06171360
Title: A Study of the Association of the Gut and Tumor Microbiome With Disease and Treatment Outcome of CDK4/6 Inhibitors in Hormone Receptor-positive HER2-negative Breast Cancer
Brief Title: A Study of the Gut Microbiome in Hormone Receptor-positive HER2-negative Breast Cancer Treated With CDK4/6 Inhibitors
Acronym: CICLIBIOME
Status: Recruiting | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/31AOU/322
Record Dates: First submitted 2023-03-13; First posted 2023-12-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal, blood and tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metastatic HR-positive HER2-negative breast cancer: Patients with metastatic HR+ HER2- BC starting a first line treatment with a CDK4/6 inhibitor (palbociclib, ribociclib, abemaciclib).
  Investigators will regularly collect blood and fecal samples for correlative translational research.
- Early HR-positive HER2-negative breast cancer at high risk of relapse: Patients with early HR+ HER2- BC at high risk of relapse, starting adjuvant treatment with a CDK4/6 inhibitor (abemaciclib, ribociclib).
  Investigators will regularly collect blood and fecal samples for correlative translational research.

SUMMARY:
Ciclibiome is a prospective study including BC patients starting treatment with a CDK4/6 inhibitor (in the metastatic and in the adjuvant setting).

This study will focus on the interplay between the gut microbiome (its composition and evolution during treatment), circulating immune, metabolic and cytokine biomarkers (before and during treatment), and response outcomes to the CDK4/6 inhibitor.

The main aim of the study is to highlight the existence of a microbial, immune and/or metabolic biomarker of response to CDK4/6 inhibition in BC, assessable by a stool or blood sample examination.

Ultimately, this will allow to study new potential combination partners for CDK4/6 inhibitors in escalation trials for poor prognosis patients.

DETAILED DESCRIPTION:
The combination of endocrine therapy and a CDK4/6 inhibitor is the preferred treatment option in advanced hormone-receptor positive (HR+) and HER2-negative (HER2-) breast cancer (BC). This combination (with abemaciclib or ribociclib) is now also considered standard of care for early HR+ HER2- BC deemed at high risk of relapse.

Biomarkers predicting response to CDK4/6 inhibition remain largely unknown. Of note, research primarily focused on acquired genomic and transcriptomic tumor cell alterations, requiring invasive biopsies of tumor content. Thus, enlarging the scope of biomarkers of response to CDK4/6 inhibition to more easily accessible biological samples and to areas other than tumoral gene pathway alterations is urgently required.

CDK4/6 inhibitors have been demonstrated to enhance the activity of cytotoxic T cells in BC, but without deep knowledge of mechanisms and implications. Studies of multiple cancer types have demonstrated the impact of the gut microbiome on the adaptive anti-cancer immunity.

Ciclibiome is a prospective study of BC patients starting treatment with a CDK4/6 inhibitor (both in the advanced and adjuvant setting), aiming to study the interplay between the gut microbiome (its composition and evolution during treatment), circulating immune, metabolic and cytokine biomarkers (before and during treatment), and response outcomes to the CDK4/6 inhibitor.

This study will explore the existence of microbial, immune and metabolic biomarkers correlated with the clinical outcomes to CDK4/6 inhibition in BC. The aim is to find an easily available biomarker, assessable by a stool or blood sample examination.

This study will generate new hypotheses, that ultimately could give rise to potential combination strategies to test in a population considered of poor prognosis.

ELIGIBILITY:
* Cohort of metastatic HR-positive HER2-negative breast cancer :

Inclusion Criteria:

Patients that respond to each of these criteria can be included :

* Diagnosis of previously untreated HR+ HER2- advanced breast cancer (defined as locally advanced and unresectable, or metastatic). HR+ defined as positive estrogen receptors as per local laboratory testing. HER2- defined as negative ISH test or an IHC status of 0 or 1+ as per local laboratory testing.
* Planned first-line treatment with an endocrine therapy (aromatase inhibitor or fulvestrant) and a CDK4/6i.
* Male or female ≥ 18 years of age at the time the informed consent is signed.
* Being able to provide written informed consent.
* Patients with a history of early breast cancer are allowed providing systemic therapy (including adjuvant endocrine therapy) was discontinued more than 6 months ago.
* Patients are willing and able to comply with the protocol for the duration of the study including sample collection.
* Paraffin-embedded tumor tissue available at diagnosis of metastatic disease (inclusion to be discussed if not available).

Exclusion Criteria:

Patients who respond to any of these criteria are excluded :

* Administration of the CDK4/6i already started.
* Concurrent or previous non breast-related malignancy in the last 3 years prior to the start of the study treatment (with the exception of a history of adequately treated cervical carcinoma in situ or non-melanoma skin cancer).
* Treatment or chronic prevention of an infection through oral or intravenous antibiotic administered less than 1 month ago. History of unique antibiotic administration as prophylaxis for an invasive procedure is allowed.
* Active disease requiring treatment with an immunomodulatory agent. Low dose oral corticosteroids (equivalent to 8 mg or less of prednisone) or topical corticosteroids are allowed.
* Serological positivity for human immunodeficiency virus (HIV) or hepatitis C (HCV).
* Known active hepatitis.
* Active inflammatory bowel disease or documented malabsorption.
* Alcohol consumption (>3 glasses/day).

  * Cohort of early HR-positive HER2-negative breast cancer at high risk of relapse :

Inclusion criteria :

Patients that respond to each of these criteria can be included :

* Early HR+ HER2- node-positive breast cancer considered at high risk of relapse (≥ 4 positive lymph nodes, or 1-3 positive lymph nodes and either or both grade 3 or tumor size > 5 cm). HR+ defined as positive estrogen receptors as per local laboratory testing. HER2- defined as negative ISH test or an IHC status of 0 or 1+ as per local laboratory testing.
* Planned adjuvant treatment with a CDK4/6i, in combination with an endocrine therapy (aromatase inhibitor or tamoxifen, with or without LHRH agonists).
* Male or female ≥ 18 years of age at the time the informed consent is signed.
* Being able to provide written informed consent.
* Patients are willing and able to comply with the protocol for the duration of the study including sample collection.
* Paraffin-embedded tumor tissue available at diagnosis of the disease or at surgical resection (inclusion to be discussed if not available).

Exclusion criteria :

Patients who respond to any of these criteria are excluded :

* Administration of the CDK4/6i already started. Ongoing administration of the endocrine therapy before study inclusion is allowed.
* Concurrent or previous non breast-related malignancy in the last 3 years prior to the start of the study treatment (with the exception of a history of adequately treated cervical carcinoma in situ or non-melanoma skin cancer).
* Treatment or chronic prevention of an infection through oral or intravenous antibiotic administered less than 1 month ago. History of unique antibiotic administration as prophylaxis for an invasive procedure is allowed.
* Active disease requiring treatment with an immunomodulatory agent. Low dose oral corticosteroids (equivalent to 8 mg or less of prednisone) or topical corticosteroids are allowed.
* Serological positivity for human immunodeficiency virus (HIV) or hepatitis C (HCV).
* Known active hepatitis.
* Active inflammatory bowel disease or documented malabsorption.
* Alcohol consumption (>3 glasses/day).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study will include HR-positive HER2-negative breast cancer patients starting treatment with a CDK4/6 inhibitor (both in the advanced and adjuvant setting).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-treatment gut microbiome composition | at study inclusion
  The pre-treatment composition of the gut microbiome is defined by 16S rRNA sequencing of the stool samples collected at study inclusion.
Pre-treatment gut metabolic profile | at study inclusion
  The pre-treatment gut metabolic profile is defined by mass spectometry on the stool samples collected at study inclusion.
Pre-treatment circulating immune population profile | at study inclusion
  The pre-treatment circulating immune population profile is defined by FACS cytometry on the blood samples collected at study inclusion.
Pre-treatment circulating metabolic profile | at study inclusion
  The pre-treatment circulating metabolic profile is defined by mass spectometry on the plasma samples collected at study inclusion.

SECONDARY OUTCOMES:
On-treatment gut microbiome composition | at 3 months, 6 months, 1 year, 2 years, 5 years
  The on-treatment composition of the gut microbiome is defined by 16S rRNA sequencing of the stool samples collected at study inclusion.
On-treatment gut metabolic profile | at 3 months, 6 months, 1 year, 2 years, 5 years
  The on-treatment gut metabolic profile is defined by mass spectometry on the stool
On-treatment circulating immune population profile | at 3 months, 6 months, 1 year, 2 years, 5 years
  The on-treatment circulating immune population profile is defined by FACS cytometry on the blood samples collected at study inclusion.
On-treatment circulating metabolic profile | at 3 months, 6 months, 1 year, 2 years, 5 years
  The on-treatment circulating metabolic profile is defined by mass spectometry on the plasma samples collected at study inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Van Marcke, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - CHU UCL Namur, Namur

IPD SHARING:
Plan to Share IPD: No